CLINICAL TRIAL: NCT00058201
Title: European Study Group For Pancreatic Cancer - Trial 3
Brief Title: Two Chemotherapy Regimens Compared With Observation in Treating Patients With Completely Resected Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Liverpool University Hospital (Other Government)
Collaborators: NCIC Clinical Trials Group (Network); Australasian Gastro-Intestinal Trials Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000287023; RLUH-NCRI-ESPAC-3V2; EU-20043; CAN-NCIC-PA2; AGITG-ESPAC-3
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-05

CONDITIONS: Pancreatic Cancer
Keywords: acinar cell adenocarcinoma of the pancreas; duct cell adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Leucovorin; Watchful Waiting

ARMS (3):
- Arm I (Active Comparator): Patients receive leucovorin calcium IV and fluorouracil IV on days 1-5.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium
- Arm II (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15.
  Interventions: Drug: gemcitabine hydrochloride
- Arm III (No Intervention): Patients undergo observation.
  Interventions: Other: clinical observation

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Arms: Arm I
Drug: gemcitabine hydrochloride — Given IV
  Arms: Arm II
Drug: leucovorin calcium — Given IV
  Arms: Arm I
Other: clinical observation — No intervention
  Arms: Arm III

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which chemotherapy regimen is more effective, or whether chemotherapy is more effective than observation, in treating pancreatic cancer after surgery.

PURPOSE: Phase III trial to compare the effectiveness of two chemotherapy regimens with no further therapy in treating patients who have completely resected pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of adjuvant gemcitabine vs fluorouracil and leucovorin calcium (vs observation only in patients with ampullary or other pancreatic malignancy), in terms of overall survival, in patients with completely resected pancreatic cancer.

Secondary

* Compare the toxicity of these regimens in these patients.
* Compare the quality of life and 5-year survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to histology (ductal adenocarcinoma vs ampullary or other pancreatic malignancy), resection margin status, and participating country. Patients are randomized to 1 of 2 treatment arms. Randomization for patients with ampullary or other pancreatic malignancy includes an observation arm.

* Arm I: Patients receive leucovorin calcium IV and fluorouracil IV on days 1-5.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15.
* Arm III (patients with ampullary or other pancreatic malignancy only): Patients undergo observation.

Treatment in arms I and II repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 3, 6, and 12 months, and then annually for 5 years.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 1,030 patients with pancreatic adenocarcinoma (515 per arms I and II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal adenocarcinoma of the pancreas OR
* Histologically confirmed diagnosis of 1 of the following types of cancer:

  * Acinar cell carcinoma or cystadenocarcinoma of the pancreas
  * Cancers of the periampullary region
  * Cancers of the intrapancreatic part of the bile duct
  * Periampullary cancers of uncertain origin
* Complete macroscopic resection (R0 or R1 resection)

  * Histological examination of all resection margins required
* No stage IVB disease
* No evidence of malignant ascites
* No liver or peritoneal metastases
* No evidence of spread to other distant abdominal or extra-abdominal organs
* No pancreatic lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* Able to participate in long-term follow-up
* No other prior or concurrent malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No serious medical or psychological condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No neoadjuvant chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* Recovered from prior resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Estimated)
Dates: Start 2001-07; Primary Completion 2008-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTC v2.0
Quality of life as measured by EORTC QLQ C-30 and ESPAC-QLQ at 3, 6, and 12 months, and then annually for 5 years
Survival rate at 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John P. Neoptolemos, MD, Study Chair — Royal Liverpool University Hospital; Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada; R. Padbury — Flinders Medical Centre; David Goldstein, MD — Institute of Oncology at Prince of Wales Hospital
Locations (27):
- Australia (2):
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
- Canada (14):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Research Institute at Queen's University, Kingston, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
- Institute for Clinical and Experimental Medicine, Preha 4, Czechia
- Tampere University Hospital, Tampere, Finland
- Hopital Tenon, Paris, France
- Universitaets-Kinderklinik Heidelberg, Heidelberg, Germany
- Agia Olga Hospital, Athens, Greece
- Petz Aladar County Hospital, Gydr, Hungary
- Policlinico Borgo Roma, Verona, Italy
- Kyoto University Hospital, Kyoto, Kyoto, Japan
- Uppsala University Hospital, Uppsala, Sweden
- Inselspital Bern, Bern, Switzerland
- Royal Liverpool University Hospital, Liverpool, England, United Kingdom

REFERENCES:
- [Result] Neoptolemos JP, Moore MJ, Cox TF, Valle JW, Palmer DH, McDonald AC, Carter R, Tebbutt NC, Dervenis C, Smith D, Glimelius B, Charnley RM, Lacaine F, Scarfe AG, Middleton MR, Anthoney A, Ghaneh P, Halloran CM, Lerch MM, Olah A, Rawcliffe CL, Verbeke CS, Campbell F, Buchler MW; European Study Group for Pancreatic Cancer. Effect of adjuvant chemotherapy with fluorouracil plus folinic acid or gemcitabine vs observation on survival in patients with resected periampullary adenocarcinoma: the ESPAC-3 periampullary cancer randomized trial. JAMA. 2012 Jul 11;308(2):147-56. doi: 10.1001/jama.2012.7352. PMID 22782416
- [Result] Neoptolemos JP, Stocken DD, Bassi C, Ghaneh P, Cunningham D, Goldstein D, Padbury R, Moore MJ, Gallinger S, Mariette C, Wente MN, Izbicki JR, Friess H, Lerch MM, Dervenis C, Olah A, Butturini G, Doi R, Lind PA, Smith D, Valle JW, Palmer DH, Buckels JA, Thompson J, McKay CJ, Rawcliffe CL, Buchler MW; European Study Group for Pancreatic Cancer. Adjuvant chemotherapy with fluorouracil plus folinic acid vs gemcitabine following pancreatic cancer resection: a randomized controlled trial. JAMA. 2010 Sep 8;304(10):1073-81. doi: 10.1001/jama.2010.1275. PMID 20823433
- [Derived] Jones RP, Psarelli EE, Jackson R, Ghaneh P, Halloran CM, Palmer DH, Campbell F, Valle JW, Faluyi O, O'Reilly DA, Cunningham D, Wadsley J, Darby S, Meyer T, Gillmore R, Anthoney A, Lind P, Glimelius B, Falk S, Izbicki JR, Middleton GW, Cummins S, Ross PJ, Wasan H, McDonald A, Crosby T, Ting Y, Patel K, Sherriff D, Soomal R, Borg D, Sothi S, Hammel P, Lerch MM, Mayerle J, Tjaden C, Strobel O, Hackert T, Buchler MW, Neoptolemos JP; European Study Group for Pancreatic Cancer. Patterns of Recurrence After Resection of Pancreatic Ductal Adenocarcinoma: A Secondary Analysis of the ESPAC-4 Randomized Adjuvant Chemotherapy Trial. JAMA Surg. 2019 Nov 1;154(11):1038-1048. doi: 10.1001/jamasurg.2019.3337. PMID 31483448
- [Derived] Ghaneh P, Kleeff J, Halloran CM, Raraty M, Jackson R, Melling J, Jones O, Palmer DH, Cox TF, Smith CJ, O'Reilly DA, Izbicki JR, Scarfe AG, Valle JW, McDonald AC, Carter R, Tebbutt NC, Goldstein D, Padbury R, Shannon J, Dervenis C, Glimelius B, Deakin M, Anthoney A, Lerch MM, Mayerle J, Olah A, Rawcliffe CL, Campbell F, Strobel O, Buchler MW, Neoptolemos JP; European Study Group for Pancreatic Cancer. The Impact of Positive Resection Margins on Survival and Recurrence Following Resection and Adjuvant Chemotherapy for Pancreatic Ductal Adenocarcinoma. Ann Surg. 2019 Mar;269(3):520-529. doi: 10.1097/SLA.0000000000002557. PMID 29068800